CLINICAL TRIAL: NCT07239960
Title: The Effect of Short-term Rhodiola Rosea Supplementation on Simulated Game Time, Perceived Fatigue, and Performance in Basketball Players
Brief Title: Short-Term Rhodiola Rosea: Effects on Hoops Players' Game Time, Fatigue & Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024219H
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Rhodiola; Sports Performance; Fatigue; Basketball Players; Exercise Physiology; Physical Performance
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, double-blind, parallel-group design. Participants are randomly assigned to either the Rhodiola supplementation group or the placebo group, and both groups receive their respective interventions simultaneously for 28 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhodiola Supplementation Group (Experimental): Participants in this arm will receive daily Rhodiola capsules for 28 days. They will undergo simulated basketball game tests and physical fitness assessments (sprint, endurance, jump tests) before and after the supplementation period.
  Interventions: Dietary Supplement: Rhodiola rosea, L
- Placebo Control Group (Placebo Comparator): Participants in this arm will receive daily placebo capsules (empty capsules identical in appearance to Rhodiola) for 28 days. They will undergo the same simulated basketball game tests and physical fitness assessments (sprint, endurance, jump tests) before and after the intervention period, without knowing their group assignment.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Rhodiola rosea, L — Participants in this arm will receive daily capsules containing Rhodiola Rosea for 28 days. The capsules are identical in appearance to placebo capsules. The intervention aims to evaluate the effects of Rhodiola supplementation on basketball players' simulated game performance, sprint times, perceived fatigue, aerobic capacity, and antioxidant markers. Participants will undergo baseline and post-intervention physical fitness assessments, including sprint tests, endurance tests, Countermovement Jump (CMJ), heart rate recovery, and simulated game tasks.
  Other Names: Golden Root, Arctic Root, R. rosea
  Arms: Rhodiola Supplementation Group
Other: Placebo Comparator — Participants in this arm will receive daily placebo capsules (identical in appearance to Rhodiola capsules) for 28 days. This group serves as a control to compare the effects of Rhodiola supplementation on basketball players' simulated game performance, sprint times, perceived fatigue, aerobic capacity, and antioxidant markers. Participants will complete the same baseline and post-intervention physical fitness assessments as the experimental group.
  Arms: Placebo Control Group

SUMMARY:
This study aims to evaluate the effects of short-term Rhodiola rosea supplementation on simulated game performance, perceived fatigue, and aerobic capacity in basketball players. The participants will include 48 professional male basketball players aged 18-25 years, all from Beijing Sport University and holding at least a national level-2 athlete certification.

The key research questions are as follows:

Does Rhodiola rosea supplementation improve the total completion time of simulated games? Does it reduce post-simulation heart rate and perceived fatigue while enhancing aerobic capacity (e.g., maximal oxygen uptake) and antioxidant indicators?

To address these questions, researchers will compare the Rhodiola rosea supplementation group (RHO group) with the control group (CTR group). Participants will be required to:

Consume Rhodiola rosea supplements or placebos (empty capsules) daily for 28 consecutive days on an empty stomach.

Complete simulated game tests-including sprints, defensive slides, and layups-with total completion time and heart rate recovery recorded.

Provide blood samples for the measurement of biochemical indicators such as total antioxidant capacity, superoxide dismutase activity, and creatine kinase.

Complete a series of physical fitness tests, including the countermovement jump (CMJ) test, 5-km run, YO-YO Intermittent Recovery Test, and maximal oxygen uptake (VO₂max) test.

DETAILED DESCRIPTION:
This study is a randomized, controlled, double-blind clinical trial aimed at evaluating the effects of short-term Rhodiola rosea supplementation on simulated game performance, perceived fatigue, physical fitness indicators, and biochemical parameters in professional basketball players. The study participants included 48 male basketball players from Beijing Sport University, all of whom were national level 2 athletes or above, ensuring a consistent training background and sports experience. The experimental design employed a strict randomization method, dividing participants into a Rhodiola rosea supplementation group (RHO group) and a control group (CTR group), with double-blind measures implemented to minimize potential bias. For example, the RHO group received a daily dose of 2.4 g of Rhodiola rosea extract (containing 0.5 g of salidroside per 100 g of raw material), while the CTR group consumed identical-looking empty capsules. All supplements were administered in a fasted state, twice daily, 30 minutes before breakfast and lunch, accompanied by an equal volume of water to control for placebo effects. Additionally, participants' daily dietary intake, including total calories, carbohydrates, proteins, and fats, was recorded throughout the study period to exclude nutritional factors as potential confounders.

In terms of experimental procedures, participants first completed baseline health assessments and physical measurements, followed by a 28-day supplementation period. Key testing sessions included simulated game testing, physical fitness tests, and blood sample collection. The simulated game test record the total time taken by participants to complete the simulated game, which includes common on-court movements such as sprints, defensive slides, and step-backs. Physical fitness tests covered multiple dimensions: the vertical jump test (CMJ) ; the YO-YO intermittent recovery test; the maximal oxygen uptake (VO₂max) test; the 5 km running test; heart rate monitoring used Polar HR monitors, with data recorded before and after tests to assess fatigue recovery.

Blood sample collection was conducted before the simulated game, with participants fasting for 8-12 hours. Venous blood samples were collected uniformly between 8:00 and 8:30 AM, followed by centrifugation to separate plasma and red blood cells, which were stored at -80°C for subsequent analysis. Biochemical indicators included plasma total antioxidant capacity (TAC) and superoxide dismutase (SOD) activity, malondialdehyde (MDA) concentration, and creatine kinase (CK) activity. Data analysis was performed using SPSS software (version 26) and GraphPad Prism (version 9.0), with continuous variables presented as mean ± standard deviation. Normality was assessed using the Shapiro-Wilk test, and a 2×2 mixed-design ANOVA [group (CTR vs. RHO) × time (pre-test vs. post-test)] was employed to evaluate intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players aged 18 years or older
* National Level 2 athletes or above with training experience
* Voluntarily participating and providing written informed consent
* Healthy, without chronic diseases, neuromuscular or musculoskeletal disorders, cardiovascular diseases, or diabetes
* Not using other nutritional supplements or alcohol-containing products during the study, and non-smokers

Exclusion Criteria:

* Allergy to Rhodiola or study-related substances
* Recent major surgery or injury affecting athletic performance
* Use of antidepressants or stimulant drugs
* Unable to comply with training or intervention requirements during the study
* Any other condition that may compromise safety or data reliability

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Total completion time of the simulated game | Baseline and after 28 days of supplementation

SECONDARY OUTCOMES:
Rating of Perceived Exertion (RPE) | Baseline and after 28 days of supplementation
Heart rate recovery | Baseline and after 28 days of supplementation
Total distance in the YO-YO intermittent recovery test | Baseline and after 28 days of supplementation
Countermovement jump (CMJ) height | Baseline and after 28 days of supplementation
Maximal oxygen uptake (VO₂max) | Baseline and after 28 days of supplementation
5 km running time | Baseline and after 28 days of supplementation
Plasma total antioxidant capacity (TAC) | Baseline and after 28 days of supplementation
Superoxide dismutase (SOD) activity | Baseline and after 28 days of supplementation
Malondialdehyde (MDA) concentration | Baseline and after 28 days of supplementation
Creatine kinase (CK) activity | Baseline and after 28 days of supplementation
BMI(kg/m^2) | Baseline and after 28 days of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from this study will be made available to other researchers for academic purposes upon reasonable request, following publication of the study results. Data sharing will comply with privacy regulations and institutional guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD) and supporting documentation will be available after publication of the study results, expected around 6 months after study completion.
Access Criteria: De-identified individual participant data (IPD) and supporting information will be available to qualified researchers upon request by contacting the corresponding author. All shared data will be de-identified to protect participant privacy, and requests will be reviewed to ensure appropriate use for academic and scientific purposes.